CLINICAL TRIAL: NCT02251678
Title: Open-Label Study to Evaluate the Effect of Elimune Capsules on Biomarkers in Patients With Plaque Psoriasis
Brief Title: Evaluate the Effect of Elimune Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elorac, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EL-1005-01-01
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-02

CONDITIONS: Plaque Psoriasis
Keywords: Plaque; Psoriasis; Biomarkers; CRP; αTNF; Interleuken
MeSH Terms: conditions — Plaque, Amyloid; Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elimune capsules (Experimental): Elimune capsules 2 capsules BID (four total capsules per day)
  Interventions: Dietary Supplement: Elimune Capsules

INTERVENTIONS:
Dietary Supplement: Elimune Capsules — 2 capsules BID for 28 days

SUMMARY:
Elorac, Inc. is evaluating the effect of Elimune™ capsules on biomarkers C-reactive protein (CRP), Tumor Necrosis Factor (αTNF), Interleuken-2 (IL-2), Interleuken-6 (IL-6), Interleuken-12 (IL-12) in subjects with plaque psoriasis with or without arthritis.

Psoriasis is a chronic inflammatory skin disease with polygenic predisposition combined with triggering factors such as trauma, inflammation or medication.

Elimune™ is a uniquely formulated prescription dietary supplement for oral administration. Each capsule contains a proprietary blend of natural ingredients, Vitamin D3, Folic Acid, Nicotinamide, Eicosapentaenoic Acid, Doscosahexaenoic Acid, Quercetin, Curcumin, Glycyrrhizin, and Hesperetin, which share anti-inflammatory activities including the ability to inhibit tumor necrosis factor-α (TNF-α).

DETAILED DESCRIPTION:
This is an open-label study consisting of a 1 day Screening Period and a 28 day Treatment Period. During the Screening Period subjects will sign informed consent and eligibility will be determined by reviewing inclusion/exclusion criteria including history of plaque psoriasis. Demographics, medical history, medication history, height and weight will be recorded. A blood sample for pre-dose biomarker analysis will be collected. Subjects will take two Elimune capsules twice daily from Day 1 to Day 28. On Day 7 and Day 28 subjects will return to the site and provide a blood sample for biomarker analysis. Adverse events and concomitant medications will be recorded throughout the study. A Physician's Evaluation of Plaque Severity and Physician's Evaluation of Arthritis Severity will be performed on Day 1, Day 7, and Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an IRB-approved informed consent prior to performing any of the screening procedures.
2. Males and females at least 18 years of age.
3. Except for plaque psoriasis with or without arthritis, subject is in generally good health.
4. Subject exhibits acutely active at least moderate to severe plaque-type psoriasis (> 5% BSA) with or without arthritis.
5. Non-pregnant, non-lactating females of childbearing potential who agree to use medically acceptable forms of birth control (abstinence, hormonal contraceptives, diaphragm with spermicide, condom with spermicide, or intrauterine device) throughout the study or females of non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or post-menopausal ≥ 1 year). A negative urine pregnancy test must be confirmed at screening for all female subjects who are not surgically sterile.
6. Non-smokers (or other nicotine use) as determined by history (no nicotine use over the past year).
7. Subject is willing and able to cooperate to the extent required by the protocol.

Exclusion Criteria:

1. Subject has known allergy or hypersensitivity to Vitamin D3, Folic Acid, Nicotinamide, Eicosapentaenoic Acid, Doscosahexaenoic Acid, Quercetin, Curcumin, Glycyrrhizin, and Hesperetin.
2. Subject has history of alcohol and/or illicit drug abuse.
3. Female subjects who are pregnant or breastfeeding.
4. History of use of any immunosuppressant products (e.g. Enbrel, Remicade, Humira) within 12 months of Day 1.
5. Use of oral corticosteroids, methotrexate, cyclosporine, ultraviolet light, or Soriatane for 90 Days prior to Day 1 and throughout the trial.
6. Use of over the counter (OTC) medications (including vitamins), prescription medications, or herbal remedies that have not been stable for 30 days prior to Day 1 or will not be stable throughout the study.
7. Use of an investigational drug within 90 days prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Individual subject serum levels of biomarkers | 28 Days
  C-reactive protein (CRP), Tumor Necrosis Factor (αTNF), Interleuken-2 (IL-2), Interleuken-6 (IL-6), and Interleuken-12 (IL-12)

SECONDARY OUTCOMES:
Physician's Evaluation of Plaque Severity | 28 Days
  Change in Physician's Evaluation of Plaque Severity from Baseline Period to Day 7 and the last day (Day 28).
Physician's Evaluation of Arthritis Severity | 28 Days
  Change in Physician's Evaluation of Arthritis Severity from Baseline Period to Day 7 and the last day (Day 28).

CONTACTS AND LOCATIONS:
Overall Officials: Scott B. Phillips, MD, Study Director — Elorac, Inc.
Locations (4):
- United States (4):
  - NMFF Dermatology Clinic, Chicago, Illinois
  - NM Lake Forest Hospital/ Women's Center, Lake Forest, Illinois
  - TKL Research, Fair Lawn, New Jersey
  - University Hospitals Case Medical Center / Dept of Dermatology, Cleveland, Ohio